CLINICAL TRIAL: NCT02723370
Title: Understanding Variability in Success of Quality Improvement for Colonoscopy
Brief Title: Implementation of Evidence Based Practices for Colonoscopy: The Strategies to Improve Colonoscopy Study
Acronym: STIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); BJC HealthCare (Other)
Responsible Party: Principal Investigator, Rebecca Lobb, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201401089; R21CA184282 (NIH)
Record Dates: First submitted 2016-03-15; First posted 2016-03-30 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Colonoscopy
Keywords: Quality of Healthcare; Colorectal neoplasms; Health Literacy; Teach-Back Communication; Evidence Based Practice; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Teach-Back Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial Intervention (Experimental): Staff will receive the intervention during the initial intervention period.
  Interventions: Behavioral: Staff multi-component implementation strategy
- Delayed Intervention (Experimental): Staff will receive the intervention during the replication study.
  Interventions: Behavioral: Staff multi-component implementation strategy

INTERVENTIONS:
Behavioral: Staff multi-component implementation strategy — Staff will receive a multi-component implementation strategy for evidence based practices (EBPs) for colonoscopy, including split-dosing of bowel preparation, low literacy education materials for patients, and teach-back procedure. The implementation strategy includes a supply of low-literacy patient education materials for split-dosing the medication of their choice, poster and pocket-card with teach-back prompts, consultation to integrate materials and teach-back into workflow and a website with additional training and patient materials.

SUMMARY:
The purpose of this study is to compare the effect of physician education about evidence based practices for colonoscopy alone, versus physician education plus a multi-component staff implementation strategy to improve adequacy of bowel preparation. Additionally the investigators will examine implementation factors that influence adoption of the evidence based practices.

DETAILED DESCRIPTION:
Over 14 million colonoscopies are performed annually in the U.S. About 25% of patients that undergo colonoscopy have inadequate bowel preparation, an impediment to identifying cancer and pre-cancerous growths. The adenoma miss rate for patients with inadequate bowel preparation can be as high as 48%. The primary goal of the Strategies to Improve Colonoscopy (STIC) study is to conduct formative research on a multi-component implementation strategy to increase staff adoption of evidence-based practices (i.e. split-dosing of the medication, low-literacy materials, teach-back) for educating patients and improving the adequacy of bowel preparation for colonoscopy.

Investigators will compare the effect of physician education about evidence based practices for colonoscopy alone, versus education plus a staff implementation toolkit to improve quality of colonoscopy (i.e. adequacy of bowel preparation). Physicians in both study groups will receive education on the evidence-based practices. Staff who work for physicians in the initial intervention group will receive a multi-component implementation strategy for the evidence-based practices, consisting of staff education, a supply of low-literacy patient education materials for split-dosing the medication of their choice, poster and pocket-card with teach-back prompts, a consultation to integrate materials and teach-back into workflow, and a website with additional training and patient materials. The initial intervention period will be followed by a replication study where the delayed intervention group will receive the intervention.

Investigators will compare change in colonoscopy quality outcomes from before to after implementation of interventions for the two study groups: a) overall; and for b) Medicaid versus other insurance using administrative and medical record data with interrupted time series analysis. Investigators will also examine factors that influence adoption of the evidence based practices using structured physician, staff and patient surveys.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who perform colonoscopies at 6 participating endoscopy centers
* Staff who work for participating physicians and provide education for bowel preparation before colonoscopy
* Patients who had an outpatient colonoscopy at a participating endoscopy center during study period

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46184 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percent of patients with adequate of bowel preparation as indicated by a Boston Bowel Preparation Scale (BBPS) score > 6 or an Aronchick scale score of fair or better. | 5 month intervention period

SECONDARY OUTCOMES:
Adoption of Evidence Based Practices | At baseline and after 5 month intervention period
  Staff report of how frequently they use the EBPs and toolkit. 5 point likert scale from 1 (Never) to 5 (Always).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Lobb, ScD, MPH, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramsey AT, Maki J, Prusaczyk B, Yan Y, Wang J, Lobb R. Using segmented regression analysis of interrupted time series data to assess colonoscopy quality outcomes of a web-enhanced implementation toolkit to support evidence-based practices for bowel preparation: a study protocol. Implement Sci. 2015 Jun 7;10:85. doi: 10.1186/s13012-015-0276-3. PMID 26050105